CLINICAL TRIAL: NCT01961115
Title: A Phase II Pilot Trial of an Indoleamine 2,3, Dioxygenase-1 (IDO1) Inhibitor (INCB024360) Plus a Multipeptide Melanoma Vaccine (MELITAC 12.1) in Patients With Advanced Melanoma
Brief Title: Epacadostat and Vaccine Therapy in Treating Patients With Stage III-IV Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Incyte Corporation (Industry); National Cancer Institute (NCI) (NIH); University of Virginia (Other)
Responsible Party: Principal Investigator, Mac Cheever, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CITN-04; NCI-2013-01605 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CITN-04 (Other: Cancer Immunotherapy Trials Network); CITN-04 (Other: CTEP); U01CA154967 (NIH)
Record Dates: First submitted 2013-10-08; First posted 2013-10-11 (Estimated); Results first posted 2018-02-07 (Actual); Last update posted 2018-06-08 (Actual); Status verified 2018-05

CONDITIONS: Mucosal Melanoma; Recurrent Melanoma; Recurrent Uveal Melanoma; Stage IIIA Skin Melanoma; Stage IIIA Uveal Melanoma; Stage IIIB Skin Melanoma; Stage IIIB Uveal Melanoma; Stage IIIC Skin Melanoma; Stage IIIC Uveal Melanoma; Stage IV Skin Melanoma; Stage IV Uveal Melanoma
MeSH Terms: conditions — Melanoma; Uveal Melanoma | interventions — epacadostat

ARMS (1):
- Treatment (epacadostat, MELITAC 12.1) (Experimental): Patients receive epacadostat PO BID on days 1-98 and receive MELITAC 12.1 peptide vaccine ID/SC on days 21, 28, 35, 56, 77, and 98 for up to 3 additional courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Epacadostat; Biological: MELITAC 12.1 Peptide Vaccine

INTERVENTIONS:
Drug: Epacadostat — Given PO
  Other Names: INCB 024360; INCB024360
Biological: MELITAC 12.1 Peptide Vaccine — Given ID/SC

SUMMARY:
This pilot phase II trial studies how well epacadostat and vaccine therapy work in treating patients with stage III-IV melanoma. Epacadostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Vaccines made from peptides and antigens may help the body build an effective immune response to kill tumor cells. Giving epacadostat with vaccine therapy may be an effective treatment for advanced melanoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the extent to which a regimen of INCB024360 (epacadostat) that normalizes serum kynurenine (Kyn)/ tryptophan (Trp) ratios alters the tumor microenvironment of melanoma, including determining the number and character of tumor-infiltrating lymphocytes as determined by examination of serial biopsies with immunohistochemistry (IHC) and gene signatures.

II. To determine the extent to which continued INCB024360 treatment plus the addition of the multipeptide melanoma vaccine, MELITAC 12.1 (MELITAC 12.1 peptide vaccine), further alters the tumor microenvironment of melanoma, including determining the number and character of tumor-infiltrating lymphocytes as determined by serial biopsies evaluating IHC and gene signatures.

SECONDARY OBJECTIVES:

I. To determine whether a regimen of INCB024360 that normalizes serum Kyn/Trp ratios plus MELITAC 12.1 vaccine changes the level or character of the vaccine-induced clusters of differentiation (CD) 8+ and CD4+ T-cell immune responses as measured in peripheral blood, as compared to prior published experience.

II. To evaluate the extent to which INCB024360 plus MELITAC 12.1 vaccine alters the number and character of peripheral blood mononuclear cell (PBMC) populations, including T and natural killer (NK) cells, as evaluated by multiparameter flow cytometry.

III. To evaluate the extent to which INCB024360 plus MELITAC 12.1 vaccine alters the PBMC transcriptome.

IV. To assess the safety and tolerability of INCB024360 plus MELITAC 12.1 vaccine.

V. To obtain preliminary data on the tumor response rate of INCB024360 plus MELITAC 12.1 vaccine by objective response rate (ORR), time to tumor progression, and overall survival.

VI. To associate any observed changes with the expression of IDO1 protein by IHC in tumor or tumor-infiltrating cells.

OUTLINE:

Patients receive epacadostat orally (PO) twice daily (BID) on days 1-98 and receive MELITAC 12.1 peptide vaccine intradermally (ID)/subcutaneously (SC) on days 21, 28, 35, 56, 77, and 98. Treatment with epacadostat may repeat every 98 days for up to 3 additional courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have malignant melanoma validated by histology or cytology; patients may have had primary cutaneous, mucosal, or ocular melanoma or metastasis from an unknown primary site

  * NOTE: patients must have measurable disease, defined as at least 1 lesion that can be accurately measured in at least 1 dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm with conventional chest x-ray or as >= 10 mm with spiral computed tomography (CT) scan, magnetic resonance imaging (MRI), or calipers by clinical exam
* Unresectable stage III or IV validated by clinical criteria (including recurrent melanoma), or patients with multiple skin/soft tissue metastases of melanoma that may be resectable but are judged to have a future recurrence risk exceeding 70% (e.g., large adenopathy, distant skin metastases or multiple in-transit melanoma metastases); tumor deemed amenable to biopsy (excisional, incisional, or core, with at least 100 mm^3 tumor volume per biopsy date) and fine-needle aspiration (FNA) biopsy

  * NOTE: optimally, patients will have tumor approachable for three serial biopsies during the trial; for patients with only one or two tumors approachable for biopsy, available tumor blocks from prior biopsies can serve as the pretreatment sample, but only if formalin-fixed tumor tissue is available and adequate to provide at least 20 unstained slides with sufficient tumor for analysis
  * NOTE: patients with unresectable advanced stage III or IV melanoma (including recurrent melanoma) are only eligible if they have failed at least one other first-line systemic therapy (other than adjuvant therapy); exceptions to this requirement are those patients who have refused and/or are ineligible for other systemic therapies
  * NOTE: v-raf murine sarcoma viral oncogene homolog B inhibitor (BRAFi) should be considered for all 'unresectable" or metastatic melanoma with BRAFV600E mutation; for low burden in-transit disease patients may enter trial without prior systemic therapy

    * Stage IV no evidence of disease (NED) is excluded by this criterion
* Patients may have had prior systemic therapy without constraint on the number of prior treatment regimens except:

  * Patients may not have had > 450 mg/m^2 doxorubicin
  * Patients may not have had > 3000 centigray (cGy) to fields encompassing the entire pelvis
* Patients must not be on any other systemic therapy within the following intervals before study enrollment:

  * 1 week after stereotactic radiosurgery of the brain or comparable technology
  * 4 weeks after cytotoxic chemotherapy or external beam radiation therapy
  * 6 weeks after chemotherapy regimens including BCNU (carmustine) or mitomycin C
  * Patients who experience melanoma progression (by Response Evaluation Criteria in Solid Tumors [RECIST] 1.1 criteria) while on or after treatment with programmed cell death 1 (PD-1) or PD ligand-1 (PDL-1) antibody may enroll on this study

    * NOTE: Patients must be off PD-1/PDL- antibody for at least 2 weeks to assess for delayed toxicity before being enrolled and receiving INCB024360; patients who are enrolled 2 weeks and up to 6 weeks after the last dose of PD-/PDL-1 antibody will enroll in cohort B and receive 100 mg BID of INCB024360; patients enrolled beyond the 6 week period after failing anti-PD-1/PDL-1 will be enrolled in cohort A; cohort A patients will receive 300 mg BID of INCB024360; patients must not have active grade 2 autoimmune toxicities attributed to these antibodies at study entry
  * 8 weeks after ipilimumab, other cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) antibody or other immunologically active antibody

    * NOTE: Patients receiving prior CTLA-4, anti-PD1 antibody or other immunologic therapy must show evidence of normal pituitary function at baseline and must not have active grade 2 autoimmune toxicities attributed to these antibodies at study entry
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1 (Karnofsky >= 70%)
* Life expectancy of at least 6 months
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 75,000/mcL
* Hemoglobin > 9 g/dL
* Total bilirubin < 1.5 x institutional upper limit of normal (bilirubin < 3 × institutional upper limit of normal for Gilbert's syndrome)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) up to 2.5 times upper limit normal (ULN)
* Creatinine < 1.5 x institutional upper limit of normal OR
* Creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Prothrombin time (PT), international normalized ratio (INR) =< 1.5 x institutional ULN unless patient is therapeutically anticoagulated; if on anticoagulants, PT/INR need to be within appropriate anticoagulation limits for the clinical indication; patients who are receiving anticoagulants may participate in the trial if their anticoagulation can be stopped safely for several days at the time of each biopsy
* Thyroid-stimulating hormone (TSH) up to 4 times ULN if thyroxine (T4) is normal
* T4 within normal limits; if abnormal and patient is receiving thyroid replacement therapy, the thyroid medication may be adjusted and the T4 may be re-tested
* Patients must express human leukocyte antigen (HLA) -A1+, -A2+, or -A3+ (80% of patients)
* Lactate dehydrogenase (LDH) < 5 × upper limits of normal

  * (NOTE: these criteria will select against patients with bulky disease and will select for patients with less disease and earlier disease)
* Participants must not have had prior autoimmune disorders requiring cytotoxic or immunosuppressive therapy, or autoimmune disorders with visceral involvement; participants must not have an active or inactive autoimmune disorders (e.g., rheumatoid arthritis, moderate or severe psoriasis, multiple sclerosis, inflammatory bowel disease, etc.); participants who are receiving therapy for an autoimmune or inflammatory disease requiring these therapies are also excluded
* The following will not be exclusionary:

  * Resolved ipilimumab associated inflammatory disease
  * The presence of laboratory evidence of autoimmune disease (e.g., positive antinuclear antibody [ANA] titer) without associated symptoms
  * Subjects with vitiligo, thyroiditis, or atopic dermatitis, but otherwise not meeting this criterion may be enrolled; individual cases can be discussed with the sponsor
* Not likely curable with surgery alone
* Not currently receiving therapy
* Females of childbearing potential must have a negative pregnancy test within 48 hours before initiating protocol therapy

  * NOTE: women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) before study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception before the study, for the duration of study participation, and 4 months after completing INCB024360 and MELITAC 12.1 administration
  * NOTE: subjects are considered not of child bearing potential if they are surgically sterile, have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy, or are postmenopausal; menopause is the age associated with complete cessation of menstrual cycles and menses, and implies the loss of reproductive potential; by a practical definition, the term assumes menopause after 1 year without menses with an appropriate clinical profile at the appropriate age
* Ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had cytotoxic chemotherapy, radiotherapy, interferon (IFN), immunosuppressive therapy, or steroids within 4 weeks (6 weeks for nitrosoureas or mitomycin C) before entering the study or those who have not recovered from adverse events (AEs) due to agents administered more than 4 weeks earlier
* Ipilimumab or other immunologically active therapy within 8 weeks of enrollment; NOTE: patients who experience melanoma progression (by RECIST 1.1 criteria) while on or after treatment with PD-1 or PDL-1 antibody may enroll on this study
* Active immunosuppressive therapy, including concurrent systemic immunosuppressive therapy or steroid therapy with more than 7 consecutive days of steroids within the prior 4 weeks

  * The use of prednisone or equivalent < 0.125 mg/kg/day (absolute maximum of 10 mg/day) as replacement therapy is permitted
  * Inhaled corticosteroids are permitted
* Cardiovascular disease that meets one of the following: congestive heart failure (New York Heart Association class III or IV), active angina pectoris, or recent myocardial infarction or acute coronary syndrome (within the last 6 months)
* History of peripheral vascular disease (PVD) that has required surgical or percutaneous intervention or documented PVD that requires medical management with medications such as acetylsalicylic acid (ASA) + clopidogrel; patients with diabetes that is not well controlled are excluded from participation; not well controlled is defined as a hemoglobin (Hgb) A1C of greater than 7.5%
* Current or history of systemic autoimmune disease requiring systemic therapy, including significant autoimmunity associated with prior ipilimumab therapy or therapy with antibodies to PD-1 or PD-L1
* Cirrhosis, chronic hepatitis C virus positivity, or chronic hepatitis B infection; subjects who may not tolerate immune-mediated hepatitis due to compromised hepatic reserve also excluded from participation including: subjects with extensive liver metastasis (as judged by the investigator); subjects who drink more than two standard alcoholic beverages per day on a regular basis; subjects who consume more than 2 grams of acetaminophen per day on a regular basis

  * A positive hepatitis B serology indicative of previous immunization (i.e., hepatitis B surface antibody [HBsAb]-positive and hepatitis B core antibody [HBcAb]-negative), or a fully resolved acute hepatitis B infection is not an exclusion criterion
* Patients who are receiving any other investigational agents for melanoma
* Patients who have had a grade one or grade two gastrointestinal adverse event during or after receiving anti-CTLA-4, anti-PD1 or anti-PD, without a colonoscopy verifying complete resolution of the adverse event
* Patients who have experienced bowel perforation, neurologic involvement, Guillain Barré syndrome, Myasthenia Gravis, Steven Johnson syndrome and other intractable events or grade 4 non-laboratory toxicity
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnancy, nursing, or unwilling to take adequate birth control during therapy

  * NOTE: pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with INCB024360 and MELITAC 12.1
* Known human immunodeficiency virus (HIV) or other history of immunodeficiency disorder

  * NOTE: HIV-positive patients taking combination antiretroviral therapy are ineligible
* Extensive active brain disease, including symptomatic brain metastases or the presence of leptomeningeal disease

  * Patients with brain metastasis, after definitive therapy with surgery or stereotactic radiation and stable off steroids for > 4 weeks, are eligible
* Any malignancy that has not been in complete remission for at least 3 years

  * NOTE: patients with cured basal or squamous cell skin cancer are not excluded; patients with a history of excised in situ cancers, including breast, cervical, colon, superficial bladder, prostate or other body system are not excluded; study entry will be allowed at the discretion of the Principal Investigator
  * NOTE: recurrence of the in situ cancer or tumor at the time of study entry would be exclusionary
* Monoamine oxidase (MAO) inhibitor use within the past 3 weeks or prior evidence of serotonin syndrome
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to INCB024360, MELITAC 12.1, or other vaccine components
* Prior organ allograft or allogeneic transplantation, if the transplanted tissue is still in place
* Medical or psychiatric illness that would, in the opinion of the investigator, preclude participation in the study or the ability of patients to provide informed consent for themselves
* History of pulmonary disease such as emphysema or chronic obstructive pulmonary disease (COPD), (forced expiratory volume in one second [FEV1] > 60% of predicted for height and age); pulmonary function tests (PFTs) are required in patients with prolonged smoking history or symptoms of respiratory dysfunction
* Use of any UDP glucuronosyltransferase 1 family, polypeptide A9 (UGT1A9) inhibitor including: acitretin, amitriptyline, androsterone, cyclosporine, dasatinib, diclofenac, diflunisal, efavirenz, erlotinib, estradiol (17-beta), flutamide, geftinib, gemfibrozil, glycyrrhetinic acid, glycyrrhizin, imatinib, imipramine, ketoconazole, lineoleic acid, mefenamic acid, mycophenolic acid, niflumic acid, nilotinib, phenobarbital, phenylbutazone, phenytoin, probenecid propofol, quinidine, ritonavir, Sorafenib, sulfinpyrazone, valproic acid and verapamil from screening through follow-up period
* Low-dose Coumadin (1 mg) is acceptable; however, doses that increase INR are not permitted; if an alternative to Coumadin-based anticoagulants cannot be used, the INR should be monitored weekly after initiation of therapy and upon discontinuation of INCB024360, until INR normalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-09-13 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2017-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Slingluff, Principal Investigator — Cancer Immunotherapy Trials Network
Locations (4):
- United States (4):
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Virginia Cancer Center, Charlottesville, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with advanced melanoma were enrolled at 4 comprehensive cancer centers in the U.S. from Sept.., 2013-Jan., 2017. Patients who failed previous standard therapies for melanoma participated in the study.
Groups:
- Cohort A: Cohort A - Pts. enrolled >6 wks after failing anti-PD-1/PDL-1 received 300 mg INCB024360 po BID every day for 98 days Cohort B - Pts. enrolled 2-6 weeks after failing anti-PD-1/PDL-1 received 100 mg INCB024360 po BID every day for 98 days All other pts. - received 300 mg po BID
  All pts received MELITAC 12.1 intradermal/subcutaneous on days 21, 28, 35, 56, 77, 98
- Cohort B: Pts. enrolled 2-6 wks after failing anti-PD-1/PDL-1 received 300 mg INCB024360 po BID every day for 98 days Cohort B - Pts. enrolled 2-6 weeks after failing anti-PD-1/PDL-1 received 100 mg INCB024360 po BID every day for 98 days
- All Other Patients: All advanced melanoma patients not previously treated with anti-PD-1 & anti-PD-L1 who meet protocol entry criteria
  Pts. will receive 300 mg INCB024360 po bid for 98 days + MELITAC 12. 1 vaccine on days 21, 28, 35, 56, 77 & 98
Period: Overall Study
Arm/Group | Cohort A | Cohort B | All Other Patients
Started | 2 | 0 | 9
Completed (The protocol called for 12 patients to be enrolled. After 3 years and 4 months only 11 pts enrolled.) | 0 | 0 | 5
Not Completed | 2 | 0 | 4
Not completed — Disease Progression | 1 | 0 | 3
Not completed — Adverse Event | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Cohort A: Pts. enrolled >6 wks after failing anti-PD-1/PDL-1 INCB024360 - 300 mg po bid continuous for 98 days MELITAC 12.1 - Intradermal/subcutaneous Days 21, 28, 35, 56, 77, 98
- Cohort B: Pts.enrolled 2-6 wks after failing anti-PD-1/PDL-1
  * INCB024360 - 100 mg po bid continuous for 98 days
  * MELITAC 12.1 - Intradermal/subcutaneous Days 21, 28, 35, 56, 77, 98
- All Other Patients: All advanced melanoma patients not previously treated with anti-PD-1 & anti-PD-L1 who meet protocol entry criteria INCB024360 - 300 mg po bid continuous for 98 days MELITAC 12.1 - Intradermal/subcutaneous Days 21, 28, 35, 56, 77, 98
- Total: Total of all reporting groups
Arm/Group | Cohort A | Cohort B | All Other Patients | Total
Number analyzed (Participants) | 2 | 0 | 9 | 11
Age, Categorical [Count of Participants; unit: Participants] — Age calculated between time of consent and date of birth.
  Participants
    <=18 years | 0 | 0 | 0 | 0
    Between 18 and 65 years | 0 | 0 | 5 | 5
    >=65 years | 2 | 0 | 4 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.5 (3.5) |  | 60.3 (14.1) | 62.2 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 5 | 6
  Male | 1 | 0 | 4 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 0 | 9 | 11
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 2 | 0 | 8 | 10
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 2 |  | 9 | 11

OUTCOME MEASURES:

1. Primary Outcome: Changes in the Concentration and Number of CD8+ Cells Infiltrating Tumor by IHC by Normalization of Kyn/Trp Ratios.
Description: Immunohistochemistry: Tumors were assessed by IHC for pattern of T-cell distribution and infiltration of cells expressing CD3 and CD8.
Time Frame: Baseline to up to day 21
Population: For one subject in cohort A day 21 tumor biopsy material was not obtained (For analysis of Cohort A n = 1). For analysis of Cohort "All Other Patients" n = 7 due to day 21 biopsy not being obtained in 2 other subjects. In addition, for one of those subjects there was no baseline tumor biopsy obtained.
Measure: Mean (Full Range); unit: Ratio: Day21CD8s/Day0CD8s
Groups:
- Cohort A: Pts.enrolled >6 wks after failing anti-PD-1/PDL-1
  Pts will receive 300mg INCB024360 p.o. bid continuous for 98 days + MELITAC 12.1 vaccine on days 21, 28, 35, 56, 77 & 98
- Cohort B: Pts.enrolled 2-6 wks after failing anti-PD-1/PDL-1
  Pts. receive 100 mg po bid INCB024360 continuous for 98 days + MELITAC 12.1 vaccine on days 21, 28, 35, 56, 77 & 98
Arm/Group | Cohort A | Cohort B | All Other Patients
Number analyzed (Participants) | 1 | 0 | 7
Ratio: Day21CD8s/Day0CD8s | 0.5 |  | 4.0 [0 to 20.2]

2. Primary Outcome: Changes in the Concentration and Number of CD8+ Cells Infiltrating Tumor by IHC by Normalization of Kyn/Trp Ratios in Combination With MELITAC 12.1
Description: Immunohistochemistry: Tumors (day 21 & day 42) were assessed by IHC for pattern of T-cell distribution and infiltration of cells expressing CD3 and CD8.
Time Frame: Day 21 up to Day 42
Population: Neither subject in cohort A had day 42 tumor biopsy material available. For analysis of Cohort "All Other Patients" n = 6 due to either a day 21 biopsy missing or a missing day 42 biopsy.
Measure: Mean (Full Range); unit: Mean Ratio: Day42CD8s/Day21CD8s
Arm/Group | Cohort A | Cohort B | All Other Patients
Number analyzed (Participants) | 0 | 0 | 6
Mean Ratio: Day42CD8s/Day21CD8s |  |  | 3.9 [0.5 to 16.8]

3. Secondary Outcome: Change in PBMC Transcriptome_v2
Description: Analysis of PBMC gene signature. This may be compared to immunologic response, tumor biopsy data and clinical response
Time Frame: Baseline to up to 16 week
Population: Data were not collected
Arm/Group | Cohort A | Cohort B | All Other Patients
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Change in the Number and Character of PBMC Populations, Including T and NK Cells, as Evaluated by Multiparameter Flow Cytometry_v2
Time Frame: Baseline to up to 1 year
Population: Data were not collected
Arm/Group | Cohort A | Cohort B | All Other Patients
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Changes in Expression of IDO1 Protein by IHC in Tumor or Tumor-infiltrating Cells_v2
Time Frame: Baseline to up to 16 weeks
Population: Data were not collected
Arm/Group | Cohort A | Cohort B | All Other Patients
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Changes in the Level or Character of the Vaccine-induced CD8+ and CD4+ Specific T-cell Immune Responses by IFN-gamma ELISPOT_v2
Description: Assessment of immunologic response will be based on a fold-increase measure from baseline as well as using a positivity threshold
Time Frame: Baseline to up to 16 weeks
Population: Data were not collected
Arm/Group | Cohort A | Cohort B | All Other Patients
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Incidence of Adverse Events Using the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0_v2
Time Frame: Up to 1 year
Population: Data were not collected
Arm/Group | Cohort A | Cohort B | All Other Patients
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Overall Response Rate Using the RECIST or Immune-Related Response Criteria (irRC)_v2
Time Frame: Up to 1 year
Population: Data were not collected
Arm/Group | Cohort A | Cohort B | All Other Patients
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Overall Survival_v2
Time Frame: From the time measurement criteria are met for complete response or partial response until the first date that recurrent and progressive disease is objectively documented, assessed up to 1 year
Population: Data were not collected
Arm/Group | Cohort A | Cohort B | All Other Patients
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Time to Tumor Progression Using RECIST or irRC_v2
Time Frame: Up to 1 year
Population: Data were not collected
Arm/Group | Cohort A | Cohort B | All Other Patients
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from initiation of therapy through study post-treatment follow-up assessments, an average of one year.
Groups:
- Cohort A: Pts. enrolled >6 wks after failing anti-PD-1/PDL-1
- Cohort B: Pts. enrolled 2-6 wks after failing anti-PD-1/PDL-1
- All Other Patients: Pts. enrolled who have not been treated with check point inhibition
  * 100 mg INCB024360 po bid continuous for 98 days
  * MELITAC 12.1 intradermal/subcutaneous on days 21, 28, 35, 56, 77, 98
  Laboratory Biomarker Analysis: Correlative studies
Arm/Group | Cohort A | Cohort B | All Other Patients
All-Cause Mortality (participants affected / at risk) | 2/2 | 0/0 | 1/9
Serious Adverse Events (participants affected / at risk) | 2/2 | 0/0 | 0/9
Other Adverse Events (participants affected / at risk) | 2/2 | 0/0 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (N=2) | Cohort B (N=0) | All Other Patients (N=9)
Ascites (Gastrointestinal disorders) | 2 (2) | 0 | 0
Syncope (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (N=2) | Cohort B (N=0) | All Other Patients (N=9)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 5 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 5 (5)
constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
injection site reaction (General disorders) | 1 (1) | 0 (0) | 9 (9)
fatigue (General disorders) | 1 (1) | 0 (0) | 4 (4)
chills (General disorders) | 0 (0) | 0 (0) | 2 (2)
flu like symptoms (General disorders) | 0 (0) | 0 (0) | 2 (2)
fever (General disorders) | 0 (0) | 0 (0) | 1 (1)
edema (General disorders) | 0 (0) | 0 (0) | 1 (1)
pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
cytokine release syndrome (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
left eyelid stye (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 2 (2)
White blood cell decreased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Investigations - Other, (Investigations) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 5 (5)
hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3)
hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
hypophospatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 3 (3)
headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
numbness in leg (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
vasovagal reaction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
skin induration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3)
pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
rash maculopapular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-27): https://cdn.clinicaltrials.gov/large-docs/15/NCT01961115/Prot_SAP_000.pdf